CLINICAL TRIAL: NCT03875547
Title: Post-marketing Surveillance (Use Result Surveillance) With Refixia®. A Multicentre, Non-interventional Post Marketing Surveillance of Safety and Effectiveness of Refixia® in Routine Clinical Care With Haemophilia B Patients in Japan.
Brief Title: Post-marketing Surveillance (Use Result Surveillance) With Refixia®
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7999-4404; U1111-1198-6270 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haemophilia B: Both patients who have not previously been exposed to Refixia® and patients previously exposed to Refixia® in one of the clinical trials can be included.
  Interventions: Drug: Refixia®

INTERVENTIONS:
Drug: Refixia® — Patients will be treated with commercially available Refixia® according to routine clinical practice at the discretion of the treating physician

SUMMARY:
The participants are invited to take part in this study because they have Haemophilia B. The purpose of this study is to assess the safety and effectiveness of Refixia® about long-term routine use in patients with Haemophilia B. The participants will get Refixia® as prescribed to them by their study doctor. The study will last up to Sep 2025 for the participant. The participants may be asked to fill in the quality of life questionnaires (if they are above age of 15). The blood samples taken from the participants as part of routine clinical practice will also be used to investigate the safety for the long-term use of Refixia®.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Refixia® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study. At each site of this study, all patients will be registered consecutively from the first patient after the launch of Refixia® (consecutively registered system).
* Diagnosis of haemophilia B in males or females, no age limitation. Patients younger than 12 years old will continue to be registered for 3 years of recruitment period regardless of the target number of patients.
* New patients who have not been previously exposed to Refixia®. Also patients previously exposed to Refixia® in NN7999-3639, -3747, -3774, -3775 or -3895 clinical trial can be enrolled in this study. The patients who have participated in NN7999 -3774 or -3895 clinical trial can be enrolled in this study as continuous cases until 30-September-2024 (one year before planned end of study date).

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Known or suspected hypersensitivity to study product or related products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia B
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Reactions (ARs) | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Count of events

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Count of events
Number of Serious Adverse Reactions (SARs) | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Count of events
Number of bleeding episodes as assessed by annualised bleeding rate (ABR) | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Count of bleeding episodes
Number of treatment requiring bleeding episodes as assessed by ABR | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Count of bleeding episodes
Haemostatic response of Refixia® in treatment of bleeds | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Haemostatic response is assessed as success/failure based on a four-point scale (excellent, good, moderate and poor) by counting excellent and good as success and moderate and poor as failure.
Haemostatic response of Refixia® in treatment of bleeds in perioperative management during surgical procedures | From baseline (week 0) to end of study (up to 6 years and 10 months)
  Haemostatic response is assessed as success/failure based on a four-point scale (excellent, good, moderate and poor) by counting excellent and good as success and moderate and poor as failure.

CONTACTS AND LOCATIONS:
Locations (23):
- Novo Nordisk Investigational Site, Søborg, Denmark
- Japan (22):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Aomori Prefectural Central Hospital_Pediatrics, Aomori
  - Matsudo City General Hospital_Pediatrics, Chiba
  - Japan Red Cross Narita Hospital_Hematology and Oncology, Chiba
  - Chiba University Hospital_Diabetes, Metabolism and Endocrinology, Chiba-shi, Chiba
  - Hyogo prefectural kobe children's hospital, Hyōgo
  - Tokyo Medical University Ibaraki Medical Center_Ibaraki, Ibaraki
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Hospital of the University of Occupational And Environmental Health Japan, Pediatrics, Kitakyusyu-shi, Fukuoka
  - Gunma University Hospital, Dept. of Hematology, Maebashi-shi, Gunma
  - Naha City Hospital_Cardiovascular Medicine, Naha-shi, Okinawa
  - Nara Medical University Hospital_Pediatrics, Nara
  - The Hospital of Hyogo College of Medicine_Haematology, Nishinomiya-shi, Hyogo
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Tokushima University Hospital_Pediatrics, Tokushima
  - Tokushima Red Cross Hospital_Pediatrics, Tokushima
  - Tokyo Medical Univ. Hospital_Laboratory Medicine, Tokyo
  - Ogikubo Hospital_Tokyo, Tokyo
  - Ishiyama Clinic, Yamagata
  - St. Marianna Univ., Yokohama City Seibu HP, Pediatrics Dept,, Yokohama-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com